CLINICAL TRIAL: NCT00211003
Title: A Multicenter, Randomized, Open-Label, Phase 3 Study to Compare the Safety and Effectiveness of Doripenem Versus a Comparator Antibiotic in Hospital-Acquired Pneumonia
Brief Title: Doripenem in the Treatment of Hospital-Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Peninsula Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005401
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Pneumonia
Keywords: Hospital-Acquired Pneumonia; Mechanical Ventilation
MeSH Terms: conditions — Pneumonia; Healthcare-Associated Pneumonia | interventions — Doripenem

INTERVENTIONS:
Drug: doripenem

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of doripenem in patients with hospital-acquired pneumonia (HAP).

DETAILED DESCRIPTION:
Doripenem is an antibiotic medication not yet approved by the US FDA. This is a phase 3, multicenter, prospective, open-label (though with blinded outcome assessments), randomized study of doripenem versus a comparator antibiotic in patients with hospital-acquired pneumonia. The study consists of screening phase, open-label treatment phase, and follow-up. Both patients on ventilator and not on ventilator are enrolled. The primary endpoint is the clinical response rate at early follow-up visit. The patients may receive either doripenem or comparator; total duration of the treatment is 7 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for >= 48 hours or those with prior hospital admission of at least 48 hours who were discharged within the last 48 hours.

Exclusion Criteria:

* Hospital-acquired pneumonia known at the time of enrollment to be caused by pathogen(s) resistant to certain antibiotics
* Any rapidly progressing disease or immediately life-threatening illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-05; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Clinical response rate at the early follow-up visit.

SECONDARY OUTCOMES:
The clinical response rate at early follow-up visit. Microbiological response rate at both early and late follow-up visits. Safety assessment (adverse events, changes in vital signs, laboratory test results) monitored throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Kollef MH, Nathwani D, Merchant S, Gast C, Quintana A, Ketter N. Medical resource utilization among patients with ventilator-associated pneumonia: pooled analysis of randomized studies of doripenem versus comparators. Crit Care. 2010;14(3):R84. doi: 10.1186/cc9012. Epub 2010 May 10. PMID 20459721
- [Derived] Kaniga K, Flamm R, Tong SY, Lee M, Friedland I, Redman R. Worldwide experience with the use of doripenem against extended-spectrum-beta-lactamase-producing and ciprofloxacin-resistant Enterobacteriaceae: analysis of six phase 3 clinical studies. Antimicrob Agents Chemother. 2010 May;54(5):2119-24. doi: 10.1128/AAC.01450-09. Epub 2010 Mar 8. PMID 20211892
- [Derived] Zhanel GG, Ketter N, Rubinstein E, Friedland I, Redman R. Overview of seizure-inducing potential of doripenem. Drug Saf. 2009;32(9):709-16. doi: 10.2165/00002018-200932090-00001. PMID 19670912
- [Derived] Rea-Neto A, Niederman M, Lobo SM, Schroeder E, Lee M, Kaniga K, Ketter N, Prokocimer P, Friedland I. Efficacy and safety of doripenem versus piperacillin/tazobactam in nosocomial pneumonia: a randomized, open-label, multicenter study. Curr Med Res Opin. 2008 Jul;24(7):2113-26. doi: 10.1185/03007990802179255. Epub 2008 Jun 11. PMID 18549664
- See also: A Multicenter, Randomized, Open-Label, Phase 3 Study to Compare the Safety and Efficacy of Intravenous Doripenem with that of Intravenous Piperacillin/Tazobactam in Hospital-Acquired Pneumonia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=641&filename=CR005401_CSR.pdf